CLINICAL TRIAL: NCT04521361
Title: Open-label, Non-randomized Phase 1, Multicenter Study to Assess Radium-223 Biodistribution in Participants With Bone Metastatic Castration Resistant Prostate Cancer (CRPC) Receiving Radium-223 Dichloride Treatment.
Brief Title: A Study to Assess How Radium-223 Distributes in the Body of Patients With Prostate Cancer Which Spread to the Bones
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20511; 2023-506435-15-00 (Registry Identifier: CTIS(EU)); 2019-000475-17 (EudraCT Number)
Record Dates: First submitted 2020-08-03; First posted 2020-08-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic castration-resistant prostate cancer (mCRPC); Single-photon emission tomography / computed tomography (SPECT/CT); radium-223,; phase I
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Low extent of disease (Experimental): Adult men with bone mCRPC having < 6 bone metastases
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Patients with High extent of disease (Experimental): Adult men with bone mCRPC having ≥ 6 bone metastases
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Drug will be administered as aqueous solution intravenously at a dose of 55 kBq/kg body weight every 4 weeks for 6 cycles (cycle length = 4 weeks).

SUMMARY:
In this study researcher want to gain more information on how the study drug (radium-223) is distributed in the bone, particularly in the tumor free bone in participants with prostate cancer. The study plans to enroll 60 patients with the age of at least 18 years and suffering from prostate cancer which has spread to the bones. Researcher will divide the study participants into 2 groups. Patients in Group 1 should have up to 6 bone metastases and patients for group 2 should have more than 6 bone metastases. The study medication will be given as injection into a vein every 4 weeks up to a maximum of 6 times. To study how radium distributes in the body and particularly in the bones, participants will undergo after study medication intake MRI or CT Scans (imaging techniques).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have histologically confirmed adenocarcinoma of the prostate.
* Participants with bone metastatic CRPC, progressing after 1 or 2 prior lines of systemic treatment for metastatic prostate cancer (including prior treatment for metastatic hormone sensitive prostate mHSPC or metastatic castration resistant prostate cancer mCRPC).
* Participants with at least 2 bone metastases on Tc 99m phosphonate whole body planar bone scans at Screening.
* Documented progression of mCRPC. Disease progression is defined by at least one of the following criteria: a. PCWG3 criteria (defined as 2 consecutive increases in PSA over a previous reference value measured at least one week prior, with a minimal start value of 1.0 ng/mL) or b. ≥2 new bone lesions (according to PCWG3 bone scan criteria) or c. Radiological progression according to RECIST, version 1.1.
* Ability to participate in the required study procedures including all scanning procedures and ability to control pain to ensure tolerance and completion of the necessary scanning procedures.
* Maintenance of medical castration or surgical castration with testosterone less than 50 ng/dL (1.7 nmol/L). If the participant is being treated with luteinizing hormone releasing hormone (LHRH) agonists or antagonists (participant who has not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to start of Screening and must be continued throughout the study.
* Participants must be on a bone health agent prior to the first dose of radium-223 dichloride. Participants with at least 6 months of prior bone health agent (BHA) treatment are preferred.
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
* Life expectancy ≥6 months.

Exclusion Criteria:

* Any chronic medical condition requiring continuous systemic corticosteroid treatment at a higher dose than 5 mg prednisone / prednisolone twice daily.
* Pathological finding consistent with neuroendocrine features small cell carcinoma of the prostate.
* Metastatic bone deposits extend of disease (EOD) grades 0 or 4 (according to centrally assessed Tc 99m phosphonate planar bone scans during Screening).
* History of visceral metastasis, or presence of visceral metastasis detected by screening imaging examinations (according to central review at screening).
* Other malignancy treated within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
* Imminent spinal cord compression based on clinical findings and / or magnetic resonance imaging (MRI). - Participants with history of spinal cord compression should have completely recovered.
* Active or symptomatic viral hepatitis
* Inability to tolerate any of the other imaging procedures in the study (ie, bone SPECT/CT and planar bone scans with a Tc 99m phosphonate radiotracer, DXA scan, radium-223 SPECT/CT scans).
* Any condition, which in the opinion of the investigator would preclude participation in this trial.
* Hypersensitivity to radium-223 dichloride.
* Blood transfusion or erythropoietin stimulating agents 4 weeks prior to start of Screening and during the whole Screening period before enrollment into the cohort.
* Prior administration of an investigational therapeutic for CRPC.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
AUC of radium-223 in tumor-free bone after 3 doses | At 4, 24 and 144 hours post injection at Cycle 3 ( total duration of one cycle is 28 days).
  The uptake of radium-223 in bone is determined with single-photon emission tomography / computed tomography (SPECT/CT).

SECONDARY OUTCOMES:
AUC of radium-223 in tumor-free bone after single dose | At 4, 24 and 144 hours post injection at Cycle 1 ( total duration of one cycle is 28 days).
AUC of radium-223 in tumor-free bone after 6 doses | At 4, 24 and 144 hours post injection at Cycle 6 ( total duration of one cycle is 28 days).

CONTACTS AND LOCATIONS:
Locations (12):
- Uniklinikum Salzburg - Landeskrankenhaus, Salzburg, Austria
- France (4):
  - ICM - Institut du Cancer de Montpellier - Val d'Aurelle, Montpellier
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancerologie Ouest - Saint-Herblain, Saint-Herblain
  - Institut Claudius Regaud - iUCT Oncopole, Toulouse
- Rambam Health Corporation, Haifa, Israel
- Azienda USL IRCCS di Reggio Emilia_Arcispedale Santa Maria Nuova - S.C. Oncologia Provinciale, Reggio Emilia, Emilia-Romagna, Italy
- Lithuania (2):
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- United Kingdom (3):
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St. Thomas' NHS Trust, St. Thomas' Hospital, London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.